CLINICAL TRIAL: NCT05790382
Title: A Phase I Study to Assess the Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Doses of NM-101 in Healthy Male and Female Subjects
Brief Title: Single and Multiple Ascending Dose Study to Assess Safety, Tolerability and Pharmacokinetics of NM-101
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Neuramedy Co. Ltd. (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NM-101-01-2022
Record Dates: First submitted 2023-03-06; First posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Parkinson Disease
Keywords: NM-101; Anti-TLR2 antibody; Blood-brain barrier; Ascending dose
MeSH Terms: conditions — Parkinson Disease | interventions — tomaralimab; rhoA GTP-Binding Protein

STUDY DESIGN:
Intervention Model Description: 56
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study. Prior to dosing visit 4 for Cohort 2, a small team will be unblinded to treatment assignment in order to conduct lumbar punctures on subjects assigned to active IMP only
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NM-101 (Experimental): Ascending doses of NM-101. IV infusion over 2 hours
  Interventions: Drug: NM-101
- Placebo (Placebo Comparator): IV infusion over 2 hours
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NM-101 — In Part 1, each cohort will receive a single dose at one of three dose levels (3 cohorts).
  In Part 2, each cohort will receive multiple doses at one of four dose levels (4 cohorts).
  Other Names: Tomarilimab; OPN-305 (formerly)
  Arms: NM-101
Drug: Placebo — Placebo solution for infusion
  Arms: Placebo

SUMMARY:
This is a Phase I, double-blind, randomised, two-part, single-ascending dose (Part 1) and multiple-ascending dose (Part 2) study of NM-101 in healthy males and healthy females of non-childbearing potential

DETAILED DESCRIPTION:
NM-101 is an anti-TLR2 antibody which may have clinical efficacy in Parkinson's disease patients. This Phase I study aims to assess the safety, tolerability and pharmacokinetics (PK) of single and multiple ascending doses of NM-101 in healthy males and healthy females of non-childbearing potential. A total of 56 subjects (8 per cohort) are planned to be enrolled.

Subjects will be randomly assigned to recieve NM-101 or placebo in a 3:1 ratio. The study will be in 2 parts: Part 1 will consist of 3 single-dose cohorts; Part 2 will consist of 4 multiple-dose cohorts.

In Part 1, sentinel dosing will be applied. In each cohort, 1 subject will be randomised to receive NM-101 and 1 subject will be randomised to receive placebo ahead of dosing in the remaining 6 subjects. The dose for Cohort 1 is 20 mg/kg NN-101. The predicted doses for Cohorts 2 and 3 are 40 mg/kg and 60 mg/kg NM-101, respectively (dependent on a blinded interim review of the safety, tolerability and PK data). Blood samples will be collected at regular intervals for PK analysis and safety from Day 1 until Day 42.

In Part 2, sentinel dosing will not be applied. Each subject will receive 4 doses of NM-101 or placebo over the course of 3 months. Dosing may occur in parallel to the conduct of Part 1. The doses administered will be selected based on emerging safety, tolerability and PK data from preceding groups in Part 1. The predicted NM-101 doses are: 10 mg/kg for Cohort 4; 20 mg/kg for Cohort 5; 40 mg/kg for Cohort 6; 60 mg/kg for Cohort 7. In Cohorts 5 to 7, subjects will undergo a lumbar puncture to assess NM-101 concentrations in the cerebrospinal fluid. Blood samples will be collected at regular intervals for PK analysis and safety from Day 1 until Day 127.

ELIGIBILITY:
Inclusion Criteria:

Informed Consent and Compliance

1. Must provide written informed consent
2. Must be willing and able to communicate and participate in the whole study

   Demographics and Contraception
3. Aged 18 to 65 years inclusive at the time of signing informed consent
4. Must agree to adhere to the contraception requirements

   Baseline Characteristics
5. Healthy males or WONCBP
6. Body mass index (BMI) of 18.0 to 32.0 kg/m2 as measured at screening

   Other
7. Must have received at least 2 doses of a COVID-19 vaccine

Exclusion Criteria:

Medical/Surgical History and Mental Health

1. Serious adverse reaction or serious hypersensitivity to any drug or formulation excipients
2. History of allergic or anaphylactic reactions to humanised or other therapeutic monoclonal antibodies or to any of the excipients of NM-101
3. Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hay fever is allowed unless it is active
4. History of clinically significant cardiovascular, renal, hepatic, dermatological, chronic respiratory or gastrointestinal disease, neurological or psychiatric disorder, as judged by the investigator
5. Undergone a lumbar puncture within 6 weeks before Day 1 (Part 2 only)
6. Medical history or evidence of mass occupying lesion in brain or spinal cord or history of spinal cord injury, which could preclude the procedure of lumbar puncture and CSF collection (Part 2 only)
7. Evidence or history of clinically significant back pain, back pathology and/or back injury (e.g. degenerative disease, spinal deformity or spinal surgery) that may predispose to complications or technical difficulties in the conduct of a lumbar puncture (Part 2 only)

   Physical Examination
8. Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator or delegate at screening

   Diagnostic Assessments
9. Evidence of current SARS-CoV-2 infection
10. History of an infection requiring treatment within 14 days of first dose of the IMP
11. A history of any ongoing, chronic or recurrent infectious disease, herpes, or evidence of tuberculosis infection as defined by a positive QuantiFERON® TB Gold test at screening
12. Clinically significant abnormal clinical chemistry, haematology or urinalysis as judged by the investigator
13. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) 1 and 2 antibody results
14. Females of childbearing potential including those who are pregnant or lactating (all female subjects must have a negative highly sensitive serum pregnancy test)

    Prior Study Participation
15. Subjects who have received any IMP in a clinical research study within the 90 days prior to Day 1, or less than 5 elimination half-lives prior to Day 1, whichever is longer
16. Subjects who have previously been administered IMP in this study. Subjects who have taken part in Part 1 are not permitted to take part in Part 2 and vice versa
17. Subjects who report to have previously received NM-101 (formerly known as OPN-305)
18. Donation of blood or plasma within the previous 3 months or loss of greater than 400 mL of blood

    Prior and Concomitant Medication
19. Subjects who are taking, or have taken, any prescribed or over-the-counter drug or herbal remedies (other than up to 4 g of paracetamol per day or HRT) in the 14 days before first IMP administration. Exceptions may apply, as determined by the investigator
20. Subjects who have had a vaccine (including COVID-19 vaccine) within 28 days before first dose
21. Have taken non-steroidal anti-inflammatory drugs or other drugs that affect coagulation or platelet function within 14 days prior to scheduled lumbar puncture (Part 2 only)

    Lifestyle Characteristics
22. History of any drug or alcohol abuse in the past 2 years
23. Regular alcohol consumption in males >21 units per week and in females >14 units per week
24. A confirmed positive alcohol breath test at screening or admission
25. Current smokers and those who have smoked within the last 12 months
26. A confirmed breath carbon monoxide reading of greater than 10 ppm at screening or admission
27. Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months
28. Confirmed positive drugs of abuse test result

    Other
29. Male subjects with pregnant or lactating partners
30. Travelled to an area where there is risk of malaria within the past year unless adequate precautions were taken
31. Subjects who are, or are immediate family members of, a study site or sponsor employee
32. Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-05-10 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-06-14 (Estimated)

PRIMARY OUTCOMES:
Safety of NM-101: Incidence of Treatment-Related Adverse Events by Severity | up to 4 months
  A treatment related adverse event is defined as a clinical event with plausible time relationship to NM-101 administration and that cannot be explained by concurrent disease or other drugs or chemicals
PK Parameter | up to 4 months
  maximum concentration (Cmax)
PK Parameter | up to 4 months
  time of the maximum measured concentration (Tmax)
PK Parameter | up to 4 months
  area under the concentration-time curve from time (AUC)
PK Parameter | up to 4 months
  First order rate constant associated with the terminal portion of the curve (Lambda-z)
PK Parameter | up to 4 months
  terminal elimination half life (t1/2)
PK Parameter | up to 4 months
  clearance (CL)
PK Parameter | up to 4 months
  Volume of distribution based on the terminal phase (Vz)
PK Parameter | up to 4 months
  Volume of distribution at steady state (Vss)

SECONDARY OUTCOMES:
Cerebrospinal Fluid (CSF) Concentrations of NM-101 | Day 2 or Day 86
  Quantification of NM-101 24 h after the dose only in Cohorts 5 to 7
Immunogenicity of NM-101 | up to 4 months
  Quantification of NM-101 anti-drug antibodies pre-dose and after each dose of NM 101
  Quantification of NM-101 anti-drug antibodies pre-dose and after each dose of NM 101 Quantification of NM-101 anti-drug antibodies pre-dose and after each dose of NM 101

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Mair, MBChB, etc., Principal Investigator — Quotient Sciences
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No